CLINICAL TRIAL: NCT04594993
Title: INFINITY™ With ADAPTIS™ Technology Total Ankle Replacement Follow-Up
Brief Title: INFINITY™ With ADAPTIS™ Technology Study
Acronym: ITAR2
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: US20-TAR-001
Record Dates: First submitted 2020-10-07; First posted 2020-10-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: INFINITY™ with ADAPTIS™ Technology Total Ankle System — Total Ankle Replacement

SUMMARY:
INFINITY™ with ADAPTIS™ Technology Total Ankle Replacement Follow-up (ITAR2) - Prospective, multi-site, multi-year post-market clinical follow-up study Study Group Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY™ Total Ankle System Number of Subjects 200 patients with up to 13 sites

DETAILED DESCRIPTION:
The selected design is a multi-center, non-randomized, prospective study of 200 subjects in the US with up to 13 investigational sites and a potential for more as needed to meet the enrollment requirements. The study subjects included are those with ankle joints damaged by severe rheumatoid arthritis, post-traumatic disease, and degenerative arthritis and implanted with the INFINITY™ With ADAPTIS™ Technology Total Ankle System.

ELIGIBILITY:
Inclusion Criteria:

* Be over 22 years of age at the time of surgery;
* Diagnosed with unilateral and/or bilateral ankle joint disease;
* Diagnosed with ankle joint damage from rheumatoid arthritis, post-traumatic, or degenerative arthritis;
* Willing and able to consent to participate (written, informed consent;
* Willing and able to attend the requested follow-up visits;
* A clinical decision has been made to use INFINITY™ with ADAPTIS™ Technology Total Ankle System replacement prior to enrollment.

Exclusion Criteria:

* Subjects with an ankle condition, as determined by the investigator, to be an inappropriate candidate for a total ankle replacement;
* Subjects requiring revision total ankle replacement of the ankle being considered for study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY™ with ADAPTIS™ Technology Total Ankle System
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2033-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Measure survivorship of INFINITY™ with ADAPTIS™ Technology Total Ankle System at 10 years | 10 years
  Assess the 10-year survivorship of 200 patients implanted with the INFINITY™ with ADAPTIS™ Technology Total Ankle System is non-inferior to other, similar devices.

SECONDARY OUTCOMES:
Radiographic Evaluation- Physician Reported Questionnaire | 10 years
  Identify and assess the implant for component loosening and/or subsidence, any radiolucency and/or cyst formation through radiographic evaluation early and throughout the lifetime of the implant.
PROMIS® Global Health Questionnaire | 10 years
  Compare the improvements in self-reported physical, mental, and social health measures from pre-op through 10 years post operatively; assessed by PROMIS® Global HealthThe PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "TScore" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Ankle Osteoarthritis Score (AOS) Questionnaire | 10 years
  Compare pain and functional improvement in the Ankle Osteoarthritis Score (AOS). AOS is a reliable, validated, visual analog-based,AOS is a reliable, validated, visual analog-based, disease-specific self-administered instrument designed specifically to measure disability and pain from ankle osteoarthritis. Both Pain and Disability components are used to calculate the total score. The score is from zero to one hundred with a lower score indicating more normal function. A minimal clinically important difference (MCID) for the Total AOS score reduction from baseline has been established: 12.35 points.
Foot & Ankle Observational Score (FAOS) questionnaire. | 10 years
  Compare the improvement in patient/physician reported function scores from pre-op through 10 years post-operatively, assessed by the Foot & Ankle Observational Score (FAOS) questionnaire. The FAOS is a self-report measure that evaluates symptoms and functional limitations in individuals with generalized foot and ankle disorders. Items for the FAOS were adapted from the Knee Injury and Osteoarthritis Outcome Score. The FAOS is composed of the following 5 subscales: pain (9 items), other symptoms (7 items), activities of daily living (7 items), sports and recreational activities (5 items), and foot and ankle-related quality of life (4 items). Each subscale has a potential range from 0 to 100. Where 100 indicates no problems and 0 indicates extreme problems.
Patient Satisfaction of Total Ankle Replacement (TAR) | 10 years
  Compare patient satisfaction of total ankle replacement (TAR) post operatively utilizing a four-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities
Locations (13):
- United States (13):
  - OrthoArizona Foot and Ankle Institute, Gilbert, Arizona
  - Eisenhower Health / Desert Orthopedic Center, Rancho Mirage, California
  - University of Colorado Orthopedic Research Center, Aurora, Colorado
  - Steadman Philippon Research Institute, Vail, Colorado
  - Florida Joint Care Institute, Trinity, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Hospital for Special Surgery, New York, New York
  - Slocum Center for Orthopedics & Sports Medicine, Eugene, Oregon
  - Southern Oregon Orthopedics, Medford, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger Institute for Clinical Research, Chattanooga, Tennessee
  - Campbell Clinic, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No